CLINICAL TRIAL: NCT01987362
Title: A Two-Part, Phase I, Multicenter, Open-Label Study of RO6870810/TEN-010 Given Subcutaneously: Part A: A Dose-Escalation Study in Patients With Advanced Solid Tumors. Part B: An Expansion Cohort in Patients With Selected Malignancies
Brief Title: A Two Part Study of RO6870810. Dose-Escalation Study in Participants With Advanced Solid Tumors and Expansion Study in Participants With Selected Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP39141; TEN-010-001 (Other: Tensha)
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumors, Advanced Solid Tumors
MeSH Terms: interventions — RO6870810

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RO6870810 (Part 1) (Experimental): Participants will receive escalated doses of RO67870810 SC. RO6870810 will be escalated at a starting dose of 0.03 milligrams per kilogram (mg/kg) to a maximum of 0.85 mg/kg. Treatment will be administered in treatment cycles of either 21 days or 28 days and continued until PD, adverse events which justify treatment withdrawal, non-adherence, non-compliance, investigator decision, lost to follow-up, enrollment in other clinical study, or unacceptable toxicity.
  Interventions: Drug: RO6870810
- RO6870810 (Part 2) (Experimental): Participants will receive RO6870810 at doses up to the MTD or up to the highest dose tested if the MTD is not defined. Treatment will be administered in treatment cycles of either 21 days or 28 days and continued until PD, adverse events which justify treatment withdrawal, non-adherence, non-compliance, investigator decision, lost to follow-up, enrollment in other clinical study, or unacceptable toxicity.
  Interventions: Drug: RO6870810

INTERVENTIONS:
Drug: RO6870810 — Participants will receive RO6870810 at different planned doses with a starting dose of 0.03 mg/kg to a maximum dose of 0.85 mg/kg SC on Days 1 to 14 in a 21-day treatment cycle or on Days 1 to 21 in a 28-day treatment cycle.
  Other Names: TEN-010

SUMMARY:
This is a Phase 1, non-randomized, dose-escalating, open label, multi-center study to be conducted in two parts (Part A and Part B). RO6870810 is a small molecule, non-covalent inhibitor of bromodomain and extra-terminal (BET) family of bromodomains. This study is designed to characterize the safety, tolerability, pharmacokinetics and anti-tumor activity of RO6870810 in participants with histologically confirmed solid tumors with progressive disease (PD) which is refractory or intolerant to standard/approved therapies. In Part A, RO6870810 will be administered by subcutaneous (SC) injection daily for either 21 consecutive days in a 28-day cycle or for 14 consecutive days in a 21-day treatment cycle in participants with advanced solid tumor malignancies to determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT). In Part B, RO6870810 will be administered at a dose up to the MTD to further characterize the safety profile and biological effect in a subset of participants with advanced solid tumor malignancies. It is anticipated that a total of 84 participants will be enrolled in to this study (54 in Part A and 30 in Part B). In addition, it is expected that up to 20 participants with histologically confirmed nuclear protein in testis (NUT)-midline carcinoma (NMC) with progressive disease requiring therapy will be enrolled in the sub-study of Parts A and B. In addition, up to 20 participants with diffuse large B-cell lymphoma (DLBCL) may be enrolled at selected study sites.

ELIGIBILITY:
Inclusion Criteria:

General:

* Participants with solid tumors must have one or more metastatic tumors evaluable or measurable on radiographic imaging
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (or 2 upon approval by the medical monitor)
* Life expectancy of greater than or equal to (>/=) 3 months
* Disease-free of active second/secondary or prior malignancies >/= 2 years with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast
* Adequate hematological, renal, hepatic and coagulation laboratory test results
* Women of child bearing potential and men must agree to use adequate contraception during the study and for 4 months after the last dose of study drug

Advanced Solid Malignancies:

* Participants with previously treated, histologically confirmed advanced solid malignancy with progressive disease requiring therapy
* Participants must be refractory or intolerant to standard therapy

NUT-midline carcinoma:

* Participants with histologically confirmed newly diagnosed or relapsed/refractory NMC with PD requiring therapy
* Diagnosis of one of the following is required:

  1. NUT Midline Carcinoma based on ectopic expression of NUT protein as determined by Immunohistochemistry (IHC) and/or;
  2. Detection of NUT gene translocation as determined by Fluorescence In-Situ Hybridization (FISH) Advanced Aggressive DLBCL
* Histologically confirmed advanced aggressive B-cell lymphoma with abnormal MYC expression with persistent disease requiring treatment
* Participants must have relapsed or progressed after at least 2 lines of prior therapy and not eligible for any curative treatment
* Participants must have measurable disease

Exclusion Criteria:

* Participants with hematologic malignancies
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia
* Have Fridericia-corrected QT interval (QTcF) greater than (>) 470 milliseconds (msec) (female) or > 450 (male), or history of congenital long QT syndrome
* Active, uncontrolled bacterial, viral, or fungal infections
* Known clinically important respiratory impairment
* Positive for human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C antibodies
* History of major organ transplant
* History of an autologous or allogeneic bone marrow transplant. For DLBCL participants only: DLBCL participants may have had a previous autologous transplant but not within 90 days of study entry
* Symptomatic central nervous system malignancy or metastasis
* Pregnant or nursing
* Treatment with surgery or chemotherapy within 28 days prior to study entry
* Prior treatment with small molecule (BET) family inhibitor
* Radiation for symptomatic lesions within 14 days of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with DLTs | Day 1 up to Day 28 (or Day 21)
MTD of RO6870810 | Day 1 up to Day 28 (or Day 21)
Percentage of Participants with Adverse Events | Baseline up to approximately 47 months

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve from Time 0 (Pre-dose) to Time 24 Hours (AUC0-24) of RO6870810 | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Pre-injection (Hour 0), immediately post-injection, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 24 and 28 hours post-injection on Day 1 Cycle 1; Pre-injection (Hour 0), immediately post-injection, 0.25, 0.5, 1, 2, and 4 hours post-injection on Day 15 Cycle 1; random samples on Days 8, 22 of Cycle 1 and on Day 1 of Cycle 2 and every cycle thereafter up to treatment completion (up to 47 months), end of treatment visit/early termination (up to 47 months) (cycle length = 21 or 28 days)
Maximum Plasma Concentration (Cmax) of RO6870810 | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Pre-injection (Hour 0), immediately post-injection, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 24 and 28 hours post-injection on Day 1 Cycle 1; Pre-injection (Hour 0), immediately post-injection, 0.25, 0.5, 1, 2, and 4 hours post-injection on Day 15 Cycle 1; random samples on Days 8, 22 of Cycle 1 and on Day 1 of Cycle 2 and every cycle thereafter up to treatment completion (up to 47 months), end of treatment visit/early termination (up to 47 months) (cycle length = 21 or 28 days)
Time to Reach Cmax (Tmax) of RO6870810 | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Pre-injection (Hour 0), immediately post-injection, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 24 and 28 hours post-injection on Day 1 Cycle 1; Pre-injection (Hour 0), immediately post-injection, 0.25, 0.5, 1, 2, and 4 hours post-injection on Day 15 Cycle 1; random samples on Days 8, 22 of Cycle 1 and on Day 1 of Cycle 2 and every cycle thereafter up to treatment completion (up to 47 months), end of treatment visit/early termination (up to 47 months) (cycle length = 21 or 28 days)
Percentage of Participants with Objective Response (Complete Response [CR] or Partial Response [PR]) Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 as Determined by the Investigator | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Screening up to PD/death whichever occurs first (assessed at screening, Day 1 of Cycle 1 and every odd numbered cycle up to treatment completion [up to 47 months], end of treatment visit [up to 47 months], and every 12 weeks thereafter up to study completion [up to 47 months]) up to 47 months (cycle length=21 or 28 days)
Median Time Taken for the First Response Based on RECIST v 1.1 as Determined by the Investigator | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Screening up to PD/death whichever occurs first (assessed at screening, Day 1 of Cycle 1 and every odd numbered cycle up to treatment completion [up to 47 months], end of treatment visit [up to 47 months], and every 12 weeks thereafter up to study completion [up to 47 months]) up to 47 months (cycle length = 21 or 28 days)
Median Time Taken for the Best Overall Response Based on RECIST v 1.1 as Determined by the Investigator | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Screening up to PD/death whichever occurs first (assessed at screening, Day 1 of Cycle 1 and every odd numbered cycle up to treatment completion [up to 47 months], end of treatment visit [up to 47 months], and every 12 weeks thereafter up to study completion [up to 47 months]) up to 47 months (cycle length = 21 or 28 days)
Progression Free Survival Based on RECIST v 1.1 as Determined by the Investigator | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Screening up to PD/death whichever occurs first (assessed at screening, Day 1 of Cycle 1 and every odd numbered cycle up to treatment completion [up to 47 months], end of treatment visit [up to 47 months], and every 12 weeks thereafter up to study completion [up to 47 months]) up to 47 months (cycle length = 21 or 28 days)
Duration of Response Based on RECIST v 1.1 as Determined by the Investigator | Baseline up to 47 months (detailed timeframe is provided in the outcome description)
  Screening up to PD/death whichever occurs first (assessed at screening, Day 1 of Cycle 1 and every odd numbered cycle up to treatment completion [up to 47 months], end of treatment visit [up to 47 months], and every 12 weeks thereafter up to study completion [up to 47 months]) up to 47 months (cycle length = 21 or 28 days)
Overall Survival | Screening up to death due to any cause (up to approximately 47 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - University Hospitals of Cleveland, Cleveland, Ohio

REFERENCES:
- [Derived] Shapiro GI, LoRusso P, Dowlati A, T Do K, Jacobson CA, Vaishampayan U, Weise A, Caimi PF, Eder JP, French CA, Labriola-Tompkins E, Boisserie F, Pierceall WE, Zhi J, Passe S, DeMario M, Kornacker M, Armand P. A Phase 1 study of RO6870810, a novel bromodomain and extra-terminal protein inhibitor, in patients with NUT carcinoma, other solid tumours, or diffuse large B-cell lymphoma. Br J Cancer. 2021 Feb;124(4):744-753. doi: 10.1038/s41416-020-01180-1. Epub 2020 Dec 14. PMID 33311588